CLINICAL TRIAL: NCT00805883
Title: MRI Targeted Focal Laser Thermal Therapy of Prostate Cancer Followed by Radical Prostatectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. John Trachtenberg, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLTT 001
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2008-12

CONDITIONS: Prostate Neoplasm
Keywords: Prostate Neoplasm; Localized; Photothermal; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: Focal Phothtermal Ablation

INTERVENTIONS:
Procedure: Focal Phothtermal Ablation — Under general anasthesia and in Lithotomy position 2-4 14 Fr laser fibers will be placed into the prostate using 3D US guidance.

SUMMARY:
This is a clinical research study designed to measure the effectiveness of focal Interstitial Laser Thermal Therapy (ILTT) at killing prostate tumours. Patients with "low risk" prostate cancer (Trans Rectal US Guided Biopsy positive) will undergo an MRI scan to try to localize the tumour. If the MRI detects the tumour they will then undergo a perineal ablative procedure (ILTT) under general anaesthetic. Seven days following ILTT they will come back to the hospital for a Radical Retoropubic Prostatectomy (RRP) procedure, which is the removal of a prostate gland through a surgical incision. After removal, the prostate will undergo further analysis to determine the exact location of cancer and evaluate the extent of cancer death caused by ILTT.

ELIGIBILITY:
Inclusion Criteria:

* Men 40-80 years of age;
* Histologically-proven prostate carcinoma;
* Prostate cancer clinical stage T1c and T2a
* Prostate MRI must confirm area suspicious for cancer in the sector of the positive biopsy;
* A minimum of six (6) weeks between the prostate biopsy and the Inclusion Visit;
* Prostate specific antigen (PSA) level 15 ng/mL

Exclusion Criteria:

* Medically unfit for Radical Retropubic Prostectomy (RRP) surgery
* Patients who are unwilling or unable to give informed consent;
* Patients with foci location in the apex of the prostate or isolated transition zone cancers
* Patients who have received androgen suppression therapy
* Patients who have received or are receiving chemotherapy for prostate carcinoma;
* Patients previously treated with surgery to the prostate (traditional, endoscopic or minimally invasive including HIFU, TUNA, RITA, microwave, TURP, cryotherapy or any curative treatment
* Patients who have undergone radiation therapy for prostate cancer or to the pelvis
* Any condition, or history of illness or surgery that, in the opinion of the Investigator, might confound the results of the study or pose additional risks to the patient (e.g. significant cardiovascular conditions or allergies);
* Patients with a history of non compliance with medical therapy and/or medical recommendations;

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Validity of MR/US Fusion and MR Targeting | 7 Days after Focal Therapy

CONTACTS AND LOCATIONS:
Overall Officials: John Trachtenberg, M.D, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lindner U, Lawrentschuk N, Weersink RA, Davidson SR, Raz O, Hlasny E, Langer DL, Gertner MR, Van der Kwast T, Haider MA, Trachtenberg J. Focal laser ablation for prostate cancer followed by radical prostatectomy: validation of focal therapy and imaging accuracy. Eur Urol. 2010 Jun;57(6):1111-4. doi: 10.1016/j.eururo.2010.03.008. Epub 2010 Mar 12. PMID 20346578
- See also: Trial Results — http://www.ncbi.nlm.nih.gov/pubmed/20346578